CLINICAL TRIAL: NCT03461224
Title: Postoperative Modulated Accelerated RAdiotherapy (MARA-1) for Early Stage Breast Cancer: a Retrospective Analysis
Brief Title: Modulated Accelerated RAdiotherapy in Early Breast Cancer
Status: Completed | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, Alessio Giuseppe Morganti, Professor, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Other Study IDs: MARA-1
Record Dates: First submitted 2018-03-05; First posted 2018-03-09 (Actual); Last update posted 2018-03-12 (Actual); Status verified 2018-03

CONDITIONS: Breast Cancer; Radiation Toxicity
Keywords: breast cancer; radiotherapy; cutaneous toxicity; subcutaneous toxicity; IMRT
MeSH Terms: conditions — Breast Neoplasms; Radiation Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MARA-1: accelerated hypofractionated RT: A forward planned IMRT technique was used and the prescribed dose to the breast was 40 Gy in 16 fx with a concomitant boost of 4 Gy.
  Interventions: Radiation: accelerated hypofractionated RT
- CG: conventional fractionated RT: In the CG, the whole breast received 50.4 Gy in 28 fractions (fx) delivered with 3D-RT, followed by a sequential boost on the tumour bed of 10 Gy in 4 fx delivered with electrons
  Interventions: Radiation: conventional fractionated RT

INTERVENTIONS:
Radiation: accelerated hypofractionated RT
  Groups: MARA-1: accelerated hypofractionated RT
Radiation: conventional fractionated RT
  Groups: CG: conventional fractionated RT

SUMMARY:
This trial was a retrospective study on postoperative accelerated hypofractionated IMRT (MARA-1) in patients with early stage breast carcinoma, to compare late toxicity after this treatment and standard fractionated RT delivered with 3D-CRT.

DETAILED DESCRIPTION:
The aim of this study was to evaluate the clinical results in terms of late skin and subcutaneous toxicity of accelerated hypofractionated forward-planned IMRT in patients with early stage BC. Results were compared with a historical control group (CG) of patients treated with 3D-conformal postoperative RT delivered with conventional fractionation.

ELIGIBILITY:
Inclusion Criteria:

* confirmed histologic evidence of pTis-pT3 breast cancer
* breast conservative surgery
* post menopausal status
* clear surgical margin

Exclusion Criteria:

* pT4
* positive or close resection margins
* 3 or more metastatic axillary nodes
* nodal irradiation
* M1

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: From 2003, all women fullfilling the inclusion criteria were treated with MARA-1 scheme
Sampling Method: Non-Probability Sample
Enrollment: 447 (Actual)
Dates: Start 2001-01-10 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-related late adverse events | 5 years
  late toxicity (cutaneous and subcutaneous) is evaluated using RTOG/EORTC criteria in both groups of patients

SECONDARY OUTCOMES:
Incidence of treatment-related acute adverse events | 6 months
  acute toxicity (cutaneous and subcutaneous) is evaluated using RTOG/EORTC criteria in both groups of patients
local control | 5 years
  absence of locoregional relapse
overall survival | 5 years
  defined as the time from diagnosis to death

CONTACTS AND LOCATIONS:
Overall Officials: Alessio G. Morganti, MD, Principal Investigator — Radiation Oncology Center, Department of Experimental, Diagnostic and Speciality Medicine-DIMES, Unversity of Bologna, S. Orsola-Malpighi Hospital, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Digesu C, Deodato F, Macchia G, Cilla S, Pieri M, Zamagni A, Farioli A, Buwenge M, Ferrandina G, Morganti AG. Hypofractionated radiotherapy after conservative surgery may increase low-intermediate grade late fibrosis in breast cancer patients. Breast Cancer (Dove Med Press). 2018 Oct 3;10:143-151. doi: 10.2147/BCTT.S167914. eCollection 2018. PMID 30323658